CLINICAL TRIAL: NCT06513299
Title: Assessing the Effectiveness of Low Tidal Volume and Low Driving Pressure in Mechanically Ventilated Severe Hypoxemic Patients: a Multicenter Emulated Target Trial
Brief Title: Effectiveness of Low Volume and Low Pressure in Severe Hypoxemic Patients
Acronym: avengARDS
Status: Active, not recruiting | Type: Observational
Sponsor: Gruppo Italiano per la Valutazione degli Interventi in Terapia Intensiva (Other)
Collaborators: Istituto Di Ricerche Farmacologiche Mario Negri (Other); University of Bari Aldo Moro (Other)
Responsible Party: Sponsor
Other Study IDs: avengARDS
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Hypoxemia; Ards
MeSH Terms: conditions — Hypoxia; Acute Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- VT1 - low tidal volume: Patients mechanically ventilated with tidal volume between 6.0 and 8.0 ml/kg PBW, until weaning conditions are satisfied. When weaning criteria are met, extubation may be attempted, it may either fail or not, or any other mechanical ventilation regime may be chosen, according to clinical practice.
  Interventions: Device: low tidal volume
- VT2 - high tidal volume: Patients mechanically ventilated with tidal volume between 8.0 and 10.0 ml/kg PBW, until weaning conditions are satisfied. When weaning criteria are met, extubation may be attempted, it may either fail or not, or any other mechanical ventilation regime may be chosen, according to clinical practice.
  Interventions: Device: high tidal volume
- ∆P1 - low driving pressure: Patients mechanically ventilated with driving pressure between 7.0 and 12.0 cmH2O, until weaning conditions are satisfied. When weaning criteria are met, extubation may be attempted, it may either fail or not, or any other mechanical ventilation regime may be chosen, according to clinical practice.
  Interventions: Device: low driving pressure
- ∆P2 - high driving pressure: Patients mechanically ventilated with driving pressure between 12.0 and 18.0 cmH2O, until weaning conditions are satisfied. When weaning criteria are met, extubation may be attempted, it may either fail or not, or any other mechanical ventilation regime may be chosen, according to clinical practice.
  Interventions: Device: high driving pressure

INTERVENTIONS:
Device: low tidal volume — Patients ventilated with assist/control modes of mechanical ventilation with tidal volume between 6.0 ml/kg PBW and 8.0 ml/kg PBW with PPLAT ≤ 30 cmH2O, until weaning criteria are met: P/F ratio > 250 mmHg; PEEP ≤ 8 cmH2O and lower than the previous day; FiO2 < 0.5 and lower than the previous day; systolic arterial pressure ≥ 85 mmHg.
  Groups: VT1 - low tidal volume
Device: high tidal volume — Patients ventilated with assist/control modes of mechanical ventilation with tidal volume between 8.0 ml/Kg PBW and 10.0 ml/kg PBW with PPLAT ≤ 30 cmH2O, until weaning criteria are met: P/F ratio > 250 mmHg; PEEP ≤ 8 cmH2O and lower than the previous day; FiO2 < 0.5 and lower than the previous day; systolic arterial pressure ≥ 85 mmHg.
  Groups: VT2 - high tidal volume
Device: low driving pressure — Patients ventilated with assist/control modes of mechanical ventilation with driving pressure between 7.0 cmH2O and 12.0 cmH2O with VT ≤ 10 ml/kg PBW, until weaning criteria are met: P/F ratio > 250 mmHg; PEEP ≤ 8 cmH2O and lower than the previous day; FiO2 < 0.5 and lower than the previous day; systolic arterial pressure ≥ 85 mmHg.
  Groups: ∆P1 - low driving pressure
Device: high driving pressure — Patients ventilated with assist/control modes of mechanical ventilation with driving pressure between 12.0 cmH2O and 18.0 cmH2O with VT ≤ 10 ml/kg PBW, until weaning criteria are met: P/F ratio > 250 mmHg; PEEP ≤ 8 cmH2O and lower than the previous day; FiO2 < 0.5 and lower than the previous day; systolic arterial pressure ≥ 85 mmHg.
  Groups: ∆P2 - high driving pressure

SUMMARY:
The present study set up to answer two questions: (a) "how low tidal volume must be to provide protective ventilatory settings able to minimize the risk of death due to Ventilator-Induced Lung Injury (VILI)?"; (b) "if protection from VILI is better achieved by targeting the driving pressure instead of the tidal volume, what is the optimal target for the driving pressure?". Solving these questions is pivotal for clinicians to personalized and precise mechanical ventilation practices to reduce the risk of VILI and avoid unnecessary risks associated to protective ventilatory settings.

Two multicenter emulated target trials will be performed using data collected with the Electronic Health Record MargheritaTre, to investigate the effect of low tidal volumes (6.0 to 8.0 ml/kg PBW vs 8.0 to 10.0 ml/kg PBW) and low driving pressures (7.0-12.0 cmH2O vs 12.0-18.0 cmH2O), respectively. Data will be used to obtain the dose-response curve of lower VT and lower ∆P in mechanically ventilated patients with acute severe hypoxemia.

ELIGIBILITY:
Inclusion Criteria:

all the following conditions present continuously for 24 hours commencing within 36 hours of ICU admission, while the patient is undergoing invasive mechanical ventilation in either flow or pressure- regulated assist/controlled modes:

1. arterial oxygen tension (PaO2) to inspiratory oxygen fraction (FiO2) ratio P/F ≤ 300 mmHg
2. hypoxemia developed within one week of a known clinical insult
3. hypoxemia not fully explained by cardiac failure or fluid overload*

Exclusion Criteria:

1. pregnancy
2. expected duration of mechanical ventilation < 48h
3. severe or moderate COPD
4. chronic liver disease
5. acute brain injury
6. patient admitted for palliative sedation
7. tumor with metastases
8. prior cardiac arrest
9. New York Heart Association Class IV
10. acute coronary syndrome
11. patients transferred from other ICUs
12. patients transferred to the ICU from the Emergency Department after a duration exceeding 24 hours in the Emergency Department
13. patients on Pressure Support Ventilation and/or patients in whom end-inspiratory plateau pressure was not measured

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted to an ICU adopting MargheritaTre as electronic health record satisfying inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 4300 (Estimated)
Dates: Start 2024-12-24 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ICU all-cause mortality | 14 days from assignment to intervention arm
  All patients will be classified as either alive if "alive at ICU discharge" or dead if "dead at ICU discharge"

SECONDARY OUTCOMES:
Ventilator-free days | 14 days from assignment to intervention arm
  Number of ventilator-free days (VFDs) during the 14 days in ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Mario Negri Institute for Pharmacological Research IRCCS, Ranica, BG, Italy

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-23): https://cdn.clinicaltrials.gov/large-docs/99/NCT06513299/Prot_SAP_002.pdf